CLINICAL TRIAL: NCT02604706
Title: RCT of Auricular Acupuncture in Substance Abuse: Effects on Anxiety, Sleep, Drug Use and Use of Addiction Treatment Services. A Randomized Controlled Study
Brief Title: Auricular Acupuncture in Substance Abuse: Effects on Anxiety, Sleep, Drug Use.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Örebro Läns Landsting (Other Government)
Responsible Party: Principal Investigator, Rickard Ahlberg, Clinical psychologist, doctoral student., Örebro Läns Landsting
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11
Record Dates: First submitted 2015-11-09; First posted 2015-11-13 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Substance Abuse; Anxiety; Sleep
MeSH Terms: conditions — Substance-Related Disorders; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NADA Acupuncture (Experimental): NADA-acupuncture was delivered in three phases: (1) one treatment each day during the first of a total of five weeks; (2) three treatments each week during the following two weeks; (3) two treatments each week during the two remaining weeks. each session consisted of approximately 40 minutes with acupuncture at five ear points called Sympathetic, Shen Men, Kidney, Liver and Lung, which are believed to be the best points for substance abuse patients. Acupuncture was administered to both ears using stainless steel needles. NADA-acupuncture were given as a supplement to treatment as usual consisting of Motivational Interview, pharmacological treatment, and control of drug use with urine tests.
  Interventions: Device: NADA Acupuncture
- LP Acupuncture (Experimental): The LP-acupuncture was delivered in two phases: (1) three treatments each week during the two first weeks; (2) two treatments each week for two weeks. each session consisted of approximately 40 minutes with acupuncture at five ear points called Sympathetic, Shen Men, Kidney, Liver and Lung, which are believed to be the best points for substance abuse patients. Acupuncture was administered to both ears using stainless steel needles. BC-acupuncture were given as a supplement to treatment as usual consisting of Motivational Interview, pharmacological treatment, and control of drug use with urine tests.
  Interventions: Device: LP acupuncture
- Relaxation (Active Comparator): Relaxation consisted of listening to soft music in a quiet room with dampened light and was delivered to match the amount and phases of the LP-acupuncture. Relaxation were given as a supplement to treatment as usual consisting of Motivational Interview, pharmacological treatment, and control of drug use with urine tests.
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Device: NADA Acupuncture — NADA-acupuncture was delivered in three phases: (1) one treatment each day during the first of a total of five weeks; (2) three treatments each week during the following two weeks; (3) two treatments each week during the two remaining weeks. each session consisted of approximately 40 minutes with acupuncture at five ear points called Sympathetic, Shen Men, Kidney, Liver and Lung, which are believed to be the best points for substance abuse patients. Acupuncture was administered to both ears using stainless steel needles. NADA-acupuncture were given as a supplement to treatment as usual consisting of Motivational Interview, pharmacological treatment, and control of drug use with urine tests.
  Arms: NADA Acupuncture
Device: LP acupuncture — The LP-acupuncture was delivered in two phases: (1) three treatments each week during the two first weeks; (2) two treatments each week for two weeks. each session consisted of approximately 40 minutes with acupuncture at five ear points called Sympathetic, Shen Men, Kidney, Liver and Lung, which are believed to be the best points for substance abuse patients. Acupuncture was administered to both ears using stainless steel needles. LP-acupuncture were given as a supplement to treatment as usual consisting of Motivational Interview, pharmacological treatment, and control of drug use with urine tests.
  Arms: LP Acupuncture
Behavioral: Relaxation — Relaxation consisted of listening to soft music in a quiet room with dampened light and was delivered to match the amount and phases of the LP-acupuncture. Relaxation were given as a supplement to treatment as usual consisting of Motivational Interview, pharmacological treatment, and control of drug use with urine tests.
  Arms: Relaxation

SUMMARY:
Background. A common alternative treatment for substance abuse is ear acupuncture. The aim of the study was to evaluate the short and long-term effect of auricular acupuncture on anxiety, sleep, drug use and addiction treatment utilization in adults with substance abuse. Method. Adults with substance abuse and psychiatric comorbidity were randomly assigned to either of two variants of auricular acupuncture - The National Acupuncture Detoxification Association protocol (NADA) or a local protocol (LP) - or relaxation training (controls). Primary outcomes were measured using the Beck Anxiety Inventory (BAI) and Insomnia Severity Index (ISI) with assessment before treatment and follow-ups after five weeks and three months. Secondary outcomes were drug use and addiction service utilization.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing patients status at the clinic.

Exclusion Criteria:

* Nickel-allergy
* Ear infection
* Heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in self rated anxiety measured with Beck Anxiety Inventory (BAI). | 5 weeks and 3 months

SECONDARY OUTCOMES:
Change in self rated sleep quality measured with Insomnia Severity Index (ISI). | 5 weeks and 3 months
Change in self rated drug use using The self-report Drug Use Disorders Identification Test (DUDIT). | 5 weeks and 3 months
Change in self rated alcohol use using The self report Alcholol Disorders Identification Test (ADUIT). | 5 weeks ans 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rickard Ahlberg, Principal Investigator — Örebro Läns Landsting
Locations (1):
- Psychiatric Research Centre, Örebro, Örebro County, Sweden

REFERENCES:
- [Derived] Ahlberg R, Skarberg K, Brus O, Kjellin L. Auricular acupuncture for substance use: a randomized controlled trial of effects on anxiety, sleep, drug use and use of addiction treatment services. Subst Abuse Treat Prev Policy. 2016 Jul 25;11(1):24. doi: 10.1186/s13011-016-0068-z. PMID 27451854